CLINICAL TRIAL: NCT00530608
Title: Electrophysiological Properties of the Pulmonary Veins
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Dr. Thomas Rostock, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: UHZ/2007/1
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2008-06

CONDITIONS: Electrophysiology of Pulmonary Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The pulmonary veins are the predominant sources of AF induction and maintenance. This study aims to assess the electrophysiological properties of the pulmonary veins and their relation to AF in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* No antiarrhythmic drug treatment
* Indication for an electrophysiological study

Exclusion Criteria:

* Structural heart diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First review of the data base with respect to study outcome was performed after 35 enrolled patients. As a result, the results were already significant and the study was stopped prematurely.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-06; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rostock, MD, Principal Investigator — University Hospital Eppendorf, Heart Center, Department of Cardiology
Locations (1):
- University Hospital Eppendorf, Heart Center, Department of Cardiology, Hamburg, Germany

REFERENCES:
- [Derived] Rostock T, Steven D, Lutomsky B, Servatius H, Drewitz I, Klemm H, Mullerleile K, Ventura R, Meinertz T, Willems S. Atrial fibrillation begets atrial fibrillation in the pulmonary veins on the impact of atrial fibrillation on the electrophysiological properties of the pulmonary veins in humans. J Am Coll Cardiol. 2008 Jun 3;51(22):2153-60. doi: 10.1016/j.jacc.2008.02.059. PMID 18510963